CLINICAL TRIAL: NCT03528278
Title: Using Motivational Techniques to Increase Levels of Physical Activity in Long Term Psychiatric Inpatient Wards
Acronym: FYSAKT
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Centre for Mental Disorders Research (NORMENT) (Unknown)
Responsible Party: Principal Investigator, Petter Andreas Ringen, Chief Consultant, Oslo University Hospital
Other Study IDs: 2012/2266
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia; Bipolar Disorder; Inpatient Facility Diagnoses; Cardiovascular Risk Factor
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Motivational Interviewing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Motivational interviewing and environmental interventions — * Revision of ward routines towards facilitating physical activity in patients and motivational work by staff
  * Education of staff with certified MI-expert organized as an intensive course and follow-up guidance. The first course held shortly before start of interventions, the rest arranged within a month
  * Training equipment
  * Motivational Interviewing (MI) techniques applied by staff
  * Weekly treatment plans including physical activity which may consist of any continuous physical exercise.

SUMMARY:
The current research project aims at investigating whether it is possible to obtain an increase in physical activity among inpatients with schizophrenia spectrum disorders by the use of motivational interviewing and environmental interventions, and whether interventions will be associated with an increase in physical fitness and/or improvement in mental health. The Norwegian health care system operates with a catchment-area based organization, which make high levels of representability of patients possible. Patients will be recruited from intermediate-long term inpatient departments where patients typically have schizophrenia spectrum disorders and are admitted for longer periods. There are thus unique possibilities for coordinated efforts to motivate for and change dysfunctional habits.

DETAILED DESCRIPTION:
The aim of the study is to investigate if motivational interviewing and environmental interventions may induce behavioral or clinical changes in intermediate-long term psychiatric in-patients with severe mental disorders.

Specific research questions:

1. Will levels of physical activity increase?
2. Will self-esteem, life satisfaction or mental or physical health improve?
3. Will it be possible to identify subgroups of patients with differentiated responses to the interventions? (i.e. for whom does it work?)

The study aims at including the majority of patients at all wards and the interventions will be additions to the ordinary treatment routines. The design is thus observational. The project will not influence the natural flow of patients through the wards during the study period. The patient population will thus be in a state of continuous change throughout the project period and the individual treatment periods will show substantial variation between patients. The total study period at one site will be 15 months. Consecutive patients will be included during a 12 month period form study start. All consenting patients admitted during this period will be assessed according to protocol at admittance and discharge, at start of interventions and every 3 months. The study will start in the first department in the first quarter of 2013 and will end in the last department the second quarter of 2015.

The main interventions will consist of change in the ward routines on several fields. The main organization of interventions will thus be according to wards and not according to individual patients as it will be difficult to direct the interventions to specific patients within the ward. As a consequence, once the interventions have started in a ward all subsequent patients admitted will necessarily receive interventions from day one of their admission into treatment.

Hypotheses will be tested by comparing assessments obtained before start of interventions with assessments obtained after a period of active interventions. As start of interventions in a ward will be an irreversible event, only patients in treatment in the ward at start of interventions will be subjects to crossover studies. Some patients will complete their treatment periods either before or after start of interventions and thus not be able to be subject to individual crossover studies. Data from these patients will be pooled in a pre-intervention and a post-intervention group respectively.

In the pre-intervention period all patients will receive individual treatment plans and make weekly plans of activity together with the staff. All patients are generally encouraged to physical training, and there are some common activities, but there is no specific focus on this. All wards have a dietary standard which include presence of fruit and raw vegetables between meals, pre-portioned dinner servings, restrictions on sugar-containing beverages and sweets and a general focus on a low-fat and high-fiber menu.

Primary measures will be measures of physical activity and fitness, clinical-physical measures or results from laboratory tests.

Procedure for informed consent and handling of data:

At start of project and at every new admittance after this point of time all patients are informed about the project and asked to give informed consent to participation. A folder is created for each individual participant (ring-binder) containing overview over assessments with time-lines and place-holders for score sheets for baseline and follow-up assessments. An information/registration sheet with the participants' signature is added to this folder.

Each unit will have a person responsible for data-collection. This person will supervise that assessments are done according to protocol, distribute registration and score sheets and collect sheets after assessments. The score sheets are added continuously to the individual folders. One person is responsible for collecting and gathering data from all units.

At the clinical wards, the project information from individuals will be stored with the same security as ordinary charts and other patient information. The research data will be put into folders which will be kept locked in a room with restricted access within the hospital premises in a 24-h locked building. Folders are only accessed when adding data (new score sheets). One person supervises this and is in charge of this local folder-database.

The contents of the score sheets are eventually punched into a central computer database with the necessary formal specifications and security measures.

Assessments at baseline only:

Diagnosis: The participants will be diagnosed with the Structural Clinical Interview for DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, version IV) for axis I disorders (SCID-I).

General and psychosocial data: Data are collected about age and gender, ethnicity, education, occupation, housing and marital/civil status.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at the psychiatric departments of Oslo University Hospital or at the Skjelfoss Psychiatric center
* DSM-IV diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, psychotic disorder not otherwise specified (NOS), bipolar I disorder or bipolar disorder NOS and/or current use of antipsychotic medication
* Informed consent to participation

Exclusion Criteria:

* Pronounced cognitive deficit (IQ < 70)
* Severe brain damage
* BMI<17.5
* Inability to speak Scandinavian or English
* Inability to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients at closed-door wards at the psychiatric departments at Gaustad and Dikemark of the Oslo University Hospital and at the Skjelfoss Psychiatric center in Hobøl.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-01-23 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2015-03-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Level of Physical Activity at 6 months | At baseline and at 6 months follow-up
  Level of physical activity is assessed by the product of the answers to the questions of frequency (range1-5), intensity (range 1-3) and duration (range 1-4) of physical activity in the Health Survey of Northern Trondelag (HUNT) questionnaire, creating a physical activity index (PA-index). A higher score indicates higher levels of activity. Total range for the PA-index is 3-60.

SECONDARY OUTCOMES:
Change from Baseline Level of Self-esteem at 6 months | At baseline and at 6 months follow-up
  Self-esteem is assessed by the Rosenberg Self-Esteem Scale. It is a ten-item Likert-type scale with items answered on a four-point scale-from strongly agree to strongly disagree. Range is 10-40.Higher values represent a better outcome.
Change from Baseline Level of Motivation at 6 months | At baseline and at 6 months follow-up
  Measures for motivation: Four visual analog scales (VAS), with range 1-10 for assessing motivation for change; self-efficacy, perceived importance, perceived obstacles/difficulty for achieving change and readiness for change. Higher values represent higher motivation.
Change from Baseline BMI at 6 months | At baseline and at 6 months follow-up
  Weight and height will be combined to report BMI in kg/m^2
Change from Baseline Life Satisfaction at 6 months | At baseline and at 6 months follow-up
  Life satisfaction is assessed by the question for life satisfaction (HUNT3 questionnaire). The range is 1-7, lower scores represent higher satisfaction.
Change from Baseline Level of Psychotic Symptoms at 6 months | At baseline and at 6 months follow-up
  The level of psychotic symptoms will be measured with The Positive and Negative Symptom Scale (PANSS), using the subscores for positive (range 7-49), negative (range 7-49) and general symptoms (range 16-112). Higher values represent a worse outcome
Change from Baseline Level of Global Symptoms (GAF-S) at 6 months | At baseline and at 6 months follow-up
  Global symptoms and psychosocial functioning are measured by the Global Assessment of Functioning Scale (GAF), the scores are split into scales of symptoms (GAF-S) and functioning (GAF-F) to improve psychometric properties. The range is from 0 (worst) to 100 (best).
Change from Baseline Level of Depressive Symptoms at 6 months | At baseline and at 6 months follow-up
  Depressive symptoms with the Montgomery Asberg Depression Rating Scale (MADRS). Range 0-60. Higher values represent a worse outcome.
Change from Baseline Level of Apathy at 6 months | At baseline and at 6 months follow-up
  Apathy is measured with the abridged 12-item (items 1,2,4,5,6,7,9,10,14,16,17,18) of the clinical version of the Apathy Evaluation Scale (AES-C-Apathy). Range 12-48. Higher values represent a worse outcome.
Change from Baseline Waist Circumference at 6 months | At baseline and at 6 months follow-up
  Waist circumference is measured with a horizontal tape measurement from the top of the right iliac crest. Measures in cm.
Change from Baseline Blood Pressure at 6 months | At baseline and at 6 months follow-up
  Systolic and diastolic blood pressure in mmHg.
Change from Baseline Blood Glucose in serum at 6 months | At baseline and at 6 months follow-up
  Glucose in serum, mmol/L
Change from Baseline HbA1C at 6 months | At baseline and at 6 months follow-up
  Glycosylated Hemoglobin (HbA1C) in full blood, %
Change from Baseline Insulin at 6 months | At baseline and at 6 months follow-up
  Insulin in serum, pmol/L
Change from Baseline Total Cholesterol at 6 months | At baseline and at 6 months follow-up
  Total Cholesterol in serum, mmol/L
Change from Baseline Triglycerides at 6 months | At baseline and at 6 months follow-up
  Triglycerides in serum, mmol/L
Change from Baseline HDL-cholesterol at 6 months | At baseline and at 6 months follow-up
  High Density Lipoprotein Cholesterol (HDL-cholesterol) in serum, mmol/L
Change from Baseline LDL-cholesterol at 6 months | At baseline and at 6 months follow-up
  Low Density Lipoprotein (LDL-cholesterol) in serum, mmol/L
Change from Baseline CRP at 6 months | At baseline and at 6 months follow-up
  C-Reactive Protein (CRP) in serum, mg/L
Change from Baseline Vitamin D at 6 months | At baseline and at 6 months follow-up
  Vitamin D total (Vit DTOT) in serum, nmol/L
Change from Baseline Level of Psychosocial Functioning (GAF-F) at 6 months | At baseline and at 6 months follow-up
  Global symptoms and psychosocial functioning are measured by the Global Assessment of Functioning Scale (GAF), the scores are split into scales of symptoms (GAF-S) and functioning (GAF-F) to improve psychometric properties. Range from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Petter Andreas Ringen, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Skjelfoss Psychiatric Centre, Hobøl
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No
Currently no IPD sharing plan

REFERENCES:
- [Derived] Ringen PA, Falk RS, Antonsen B, Faerden A, Mamen A, Rognli EB, Solberg DK, Martinsen EW, Andreassen OA. Using motivational techniques to reduce cardiometabolic risk factors in long term psychiatric inpatients: a naturalistic interventional study. BMC Psychiatry. 2018 Aug 15;18(1):255. doi: 10.1186/s12888-018-1832-6. PMID 30111298